CLINICAL TRIAL: NCT06190054
Title: Evaluation of the Efficacy and Safety of an Eye Drops With Hydroxypropyl-methylcellulose and Inositol as Principal Components (MERAMIRT®) in the Treatment of Dry Eye Disease Associated to Asthenopia and Accommodative Effort in Video Display Terminal Users
Brief Title: Evaluation of Performance and Safety of Eye Drops With Hydroxypropyl-methylcellulose and Inositol in Drye Eye Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IS44-21-01
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2023-12

CONDITIONS: Dry Eye Disease Associated to Asthenopia and Accommodative Effort in Video Display Terminal Users

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MERAMIRT (Experimental): Patients with diagnosis of moderate to severe dry eye disease with asthenopia and accommodative effort will receive MERAMIRT®, 1-2 drop per eye 3 times a day for 90 days.
  Interventions: Device: MERAMIRT

INTERVENTIONS:
Device: MERAMIRT — MERAMIRT®, a class IIa medical device, is indicated for hydration and lubrication of the ocular surface under conditions of eye disorders caused by environmental, visual and mechanical stress, also due to asthenopia and accommodation effort. The main component of MERAMIRT® are Hydroxypropyl-methylcellulose (HPMC 0.3%) and Inositol (0.1%).
  HPMC has the property of moisturizing and lubricating the eye. Inositol is used with an antioxidant role

SUMMARY:
This is a profit, multicentric, prospective, single-arm, open-label, non-pharmacological clinical investigation.

Patients with diagnosis of moderate to severe dry eye disease with asthenopia and accommodative effort will receive MERAMIRT®, 1-2 drop per eye 3 times a day for 90 days.

DETAILED DESCRIPTION:
MERAMIRT®, a class IIa medical device, is indicated for hydration and lubrication of the ocular surface under conditions of eye disorders caused by environmental, visual and mechanical stress, also due to asthenopia and accommodation effort. The main component of MERAMIRT® are Hydroxypropyl-methylcellulose (HPMC 0.3%) and Inositol (0.1%).

HPMC has the property of moisturizing and lubricating the eye. Inositol is used with an antioxidant role.

Hypromellose is a polymer that has the property to tick and stabilize the tear film on the corneal surface, which create a protective, transparent and viscoelastic layer. Inositol, as other osmolytes, may contribute to counteract the oxidant action on free radicals produced in condition of asthenopia and accommodative effort. Such activity may indirectly support the muscular metabolic processes favoring the contractile response.

MERAMIRT® is a hydrating and lubricant tear replacement indicated in ocular isturbances caused by environmental, visual and mechanic stress, also due to asthenopia and accommodative effort.

In a small, open-label study, a 0.3% hypromellose eye gel showed statistically significant effects in relieving ocular symptoms and in improving ocular comfort in patients with dry eye syndrome.

Another recent study showed that treatment with punctual occlusion using hypromellose 2% was associated with a significant reduction in signs and symptoms in patients with dry eye.

Based on the preliminary available background on the use of hypromellose in the management of dry eye syndrome, this investigation has been designed to assess the efficacy and safety of a sterile ophthalmic solution that contains hypromellose and inositol (MERAMIRT®), in a sample of VDT users suffering of moderate or severe DED with asthenopia and accommodative effort.

ELIGIBILITY:
Inclusion Criteria:

1. Patients having signed written informed consent to participate in the study obtained according to Good Clinical Practice (GCP);
2. Patients having an age ≥ 18 years;
3. Patients with a diagnosis of moderate or severe dry eye disease (according to TFOS DEWS II definition) with asthenopia and accommodative effort, assessed through the following exams: visual acuity, intraocular pressure, slit lamp examination, Schirmer's test, TBUT, corneal and conjunctival staining (Oxford Staining Scheme), CVS-Q and SPEED questionnaires or previous diagnosis of dry eye disease not treated in the previous 15 days;
4. Schirmer's test ≤ 10 mm;
5. TBUT ≤ 10 sec;
6. Fluorescein staining of the cornea and conjunctiva (Oxford scale value ≤ 2); In case of bilateral dry eye syndrome, only the worst eye, defined as the eye with the higher severity of impairment according to the Investigator's judgment based on the above exams, will be considered for assessments (although both eyes will be treated). In the case of bilateral dry eye syndrome with both eyes having the same level of impairment, the right eye will be considered for assessments by convention.
7. Use of video terminal display more than 4 hours daily, at least five days per week (minimum twenty hours a week);
8. Patients being able to comprehend the full nature and the purpose of the investigation, including possible risks and side effects, and subjects able to cooperate with the Investigator and to comply with the requirements of the entire investigation (including ability to attend all the planned study visits according to the time limits), based on Investigator's judgment;
9. Patients agree to not apply during the study any other eye drops product that could interfere (particularly, corticosteroid and antibiotics eye drops) with the investigational product. Use of contact lenses during then study is permitted, but they are to be removed in the 24 hours preceding each visit and prior each MERAMIRT® application;
10. Female patients having a negative urine pregnancy test result at screening and using an appropriate method of contraception for at least 30 days before inclusion and during the whole investigation period, according to the definition of Note 3 of ICH M3 Guideline*, if females of childbearing potential (i.e., not permanently sterilized - post hysterectomy or tubal ligation status - or not postmenopausal):

    * Note: According to the definition of Note 3 of ICH M3 Guideline a highly effective method is defined as those which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly.Highly effective birth control methods include: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable); intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomised partner; sexual abstinence.

Exclusion Criteria:

1. Patients under treatment with any therapy (drug, medical device or any other eye drops product, particularly, corticosteroid and antibiotics eye drops) that could interfere with the assessment of the efficacy or incidence of adverse events;
2. Patients with presence or history of any systemic or ocular disorder, condition or disease (with particular attention to malignancies and neuro-oncological diseases) that, according to Investigator's judgment, can interfere with the conduct of the required investigation procedures or the assessment of the efficacy or the interpretation of the investigation results or the incidence of adverse events;
3. Patients suffering from diseases or conditions that could interfere with the assessment of the efficacy or incidence of adverse events, such as uncorrected presbyopia, myopia astigmatism, hyperopia;
4. Patients with hypersensitivity and/or allergy to any of the MERAMIRT® ingredients;
5. Patients not giving their written informed consent;
6. Patients not being able to apply during the study any eye drops product;
7. Patients participating to another clinical study/investigation at the same time as the present investigation or within 30 days;
8. Patients who have history of drug, medication or alcohol abuse or addiction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy Assessment of dry eye symptoms from baseline | Day 30
  Change from baseline in TBUT value. The TBUT will be measured twice during the first minute after the instillation of the fluorescein. If the 2 readings differ by more than 2 seconds a third reading will be taken. The TBUT value will be the average of the 2 or 3 measurements

SECONDARY OUTCOMES:
Efficacy Assessment of dry eye symptoms from baseline | Day 30 and Day 60
  Change from baseline in TBUT value. The TBUT will be measured twice during the first minute after the instillation of the fluorescein. If the 2 readings differ by more than 2 seconds a third reading will be taken. The TBUT value will be the average of the 2 or 3 measurements
Assessment of ocular surface health from baseline | Day 30, Day 60 and Day 90
  Change from baseline of the quality of the cornea and the conjunctiva, as measured using the Oxford Grading Scale using the fluorescein staining test.
  Corneal and conjunctival staining will be conducted using fluorescein instillation into the tear film, and the score will be measured using the Oxford grading scheme. The degree of staining will be based on the number of dots on a series of six panels (A-E). In each panel, fluorescein staining is represented by punctate dots and the staining score will range from 0 to 5 for each panel, for a total possible score ranging from 0 to 15 for the exposed interpalpebral conjunctiva and cornea (Bron et al, 2003). Specifically, the keratoconjunctival staining will be rated mild (stage 0 or 1), moderate (stage 2 or 3), or severe (stage 4 or 5).
Efficacy Assesment of drye eye symptoms in visual-related function from baseline | Day 30, Day 60 and Day 90
  Change from baseline in computer-vision syndrome questionnaire (CVS-Q) scores. The CVS-Q questionnaire will be used to measure the following symptoms of CVS: eye fatigue, headache, blurred vision, double vision, itching eyes, dryness, tearing, eye redness and pain, excessive blinking, feeling of a foreign body, burning or irritation, difficulty in focusing for near vision, feeling of sight worsening, and sensitivity to light (Gonzalez-Perez et al, 2014). The CVS-Q questionnaire measures the frequency of the above-mentioned symptoms with the response options of "never," "occasionally," and "often or always." If the participants report to have symptoms "occasionally," or "often," they will be asked to rate the intensity of the symptoms, choosing between the options "moderate" or "intense."
Efficacy Assessment of patient-subjective evaluation of ocular symptoms from baseline | Day 90
  Change from baseline in Standardized Patient Evaluation of Eye Dryness (SPEED)questionnaire scores.
  The Standardized Patient Evaluation of Eye Dryness (SPEED) questionnaire gives a score from 0 to 28 that is the result of 8 items that assess frequency and severity of symptoms (Ngo et al, 2013). The symptoms assessed include dryness, grittiness, scratchiness, irritation, burning, watering, soreness, and eye fatigue. The questionnaire assesses whether these symptoms were not problematic (score 0), tolerable (score 1), uncomfortable (score 2), bothersome (score 3), or intolerable (score 4)
Efficacy Assessment of visual acuity from baseline | Day 90
  Visual function will be assessed by distance visual acuity measurement measured with the Snellen chart, uncorrected distance visual acuity (UDVA, vision with no extraocular optical correction) and best corrected distance visual acuity (BCVA, defined as obtained with the best possible refractive correction). Visual acuity values will be expressed in decimal, fraction or logMAR. All assessments will be performed using standard charts and procedures at specified visual angle, illumination and contrast. Current refraction will be determined prior to visual acuity testing to obtain best-corrected vision.
Assessment of of patients' production of aqueous tears from baseline | Day 30, Day 60 and Day 90
  Change from baseline the Schirmer's test I values. The Schirmer's test I is one of the commonly used methods to assess the aqueous tear production. A paper strip is inserted into the eye, under the eyelid, in the lower fornix near the lateral corner, away from the cornea, for five minutes to measure the production of tears. The wet portion of the strip is measured in millimeters. Values above 10 mm have to be considered normal
Assessment of Incidence and nature of Adverse Effects | Day 90
  Incidence and nature of the Serious Adverse Device Effects (SADEs); Incidence and nature of the Adverse Device Effects (ADEs); Incidence and nature of Investigational Medical Device Deficiencies (IMDDs).

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Rosa, MD, Principal Investigator — AOU-San Giovanni di Dio e Ruggi d'Aragona- Salerno
Locations (4):
- Italy (4):
  - ASST Bergamo Est-Ospedale M.O.A. Locatelli, Piario, Bergamo
  - Fondazione Policlinico Universitario Campus Biomedico, Roma, RO
  - AOU- San Giovanni di Dio e Ruggi d'Aragona, Salerno
  - Ospedale Bel Colle, Viterbo

IPD SHARING:
Plan to Share IPD: No